CLINICAL TRIAL: NCT04745546
Title: Guo's Visceral Arteries Reconstruction: The First in Man Study of WeFlow-JAAA Stent Graft System
Brief Title: Guo's Visceral Arteries Reconstruction :The First in Man Study of WeFlow-JAAA Stent Graft System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Endonom Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WeFlow-JAAA V1.0
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Juxta Renal Abdominal Aortic Aneurysm Without Rupture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WeFlow-JAAA Stent Graft System (Experimental): Participants will be treated with WeFlow-JAAA Stent Graft System
  Interventions: Device: WeFlow-JAAA Stent Graft System

INTERVENTIONS:
Device: WeFlow-JAAA Stent Graft System — The abdominal aorta stent graft system consists of the abdominal aorta embedded stent system, the abdominal aorta bifurcation stent system and the extended stent system. The abdominal aorta embedded stent has two embedded branch stents and two fenestrations. It can be combined with a peripheral small stent system of appropriate specifications to reconstruct the superior mesenteric artery, bilateral renal arteries and keep the abdominal trunk unobstructed. At the same time, the combination of the abdominal aorta embedded stent, the abdominal aorta bifurcation stent and the extended stent can solve the proximal renal and transrenal abdominal aortic aneurysm lesions with the upper edge of the abdominal aortic aneurysm body and the lower edge of the superior mesenteric artery opening ≥ 5 mm.

SUMMARY:
This study is the First in Man Study of WeFlow-JAAA Stent Graft System manufactured by EndoNom Medtech(Hangzhou) Co., Ltd.

DETAILED DESCRIPTION:
This clinical trial was conducted in a qualified clinical trial institution. Investigators will use WeFlow-JAAA Stent Graft System manufactured by EndoNom Medtech (Hangzhou) Co., Ltd. to treat patients with juxta renal abdominal aortic aneurysms. This is a Prospective, single-center, first in man study to evaluate the safety and effectiveness of abdominal aorta stent graft system in the treatment of patients with juxta renal abdominal aortic aneurysms. Follow-up will be conducted before discharge, 30 days after surgery, 6 months after surgery and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1.18 to 80 years old； 2.Able to understand the purpose of the trial, participate in the trial voluntarily with informed consent form signed by the patient him/herself or his or her legal representative, and willing to complete follow-up visits as required under the protocol; 3.Diagnosed as a perirenal abdominal aortic aneurysm, and need to reconstruct the superior mesenteric artery and both renal arteries blood supply； 4.The diameter of the proximal anchoring area (abdominal aorta at the lower edge of the superior mesenteric artery opening) is 18-34mm； 5.The upper edge of the aneurysmal body is more than 5mm from the lower edge of the superior mesenteric artery opening； 6.The distance between the bifurcation of the renal artery and the opening of the renal artery is more than 15mm, and the diameter range of the beginning of the renal artery is 5-8mm； 7.The twist angle of the proximal tumor neck (the angle between the long axis of the normal abdominal aorta and the long axis of the tumor neck) ≥120°； 8.With proper femoral artery, iliac artery, and brachial artery approach, aortic endovascular treatment can be performed.

Exclusion Criteria:

1. Severe stenosis, calcification and mural thrombosis in the proximal anchoring area；
2. Pregnant, breastfeeding or cannot contraception during the trial period;
3. The patient has participated in clinical trials of other drugs or devices during the same period；
4. Need to intervene in other vascular diseases (such as coronary artery and carotid artery) during the same operation and the postoperative drug treatment plan is affected；
5. Have history of aortic surgery or endovascular repair surgery；
6. Allergic to contrast agents, anesthetics, stents and delivery materials；
7. Cannot tolerate anesthesia；
8. Severe liver, kidney, lung, and heart function abnormalities before surgery [Serum creatinine exceeds 2 times the upper limit of normal; alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeds 5 times the upper limit of normal ;Serum total bilirubin (STB) more than 2 times the upper limit of normal; Left ventricular ejection fraction is lower than normal by cardiac color Doppler ultrasound examination]；
9. Ruptured abdominal aortic aneurysm, pseudo aortic aneurysm and dissecting aortic aneurysm；
10. History of myocardial infarction, TIA or cerebral infarction within the past 3 months；
11. Contraindications in the treatment of antiplatelet agents and anticoagulants；
12. Life expectancy is less than 12 months (such as advanced malignant tumors)
13. Acute systemic infection
14. Investigator judged that not suitable for interventional treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoint | 30 days
  No major adverse events related to device or surgery within 30 days after surgery :
  Major adverse events within 30 days after surgery are all-cause death, myocardial infarction, renal failure, respiratory failure, ischemic stroke, intestinal necrosis, severe ischemia, or necrosis of lower limbs.
Primary effective endpoint | 12 months
  Treatment success rate of abdominal aortic aneurysm 12 months after operation.

SECONDARY OUTCOMES:
Secondary safety endpoint | 30 days, 6 months, 12 months
  All-cause mortality, abdominal aortic aneurysm-related mortality, serious adverse events, device-related adverse events:
  1. All-cause mortality 30 days, 6 months, 12 months after operation.
  2. Abdominal aortic aneurysm related mortality 30 days, 6 months, 12 months after operation.
  3. The incidence of serious adverse events 30 days, 6 months, 12 months after operation.
  4. The incidence of device-related adverse events 30 days, 6 months, 12 months after operation.
Secondary effective endpoint | 30 days, 6 months, 12 months
  The incidence of type I or type III endoleak, the incidence of stent graft displacement, the patency rate of branch vessels, the incidence of conversion to open surgery or secondary interventional surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao JP, Zhang HP, Xiong J, Jia X, Ma XH, Wang LJ, Xu YL, Zhang MH, Guo W. First-in-Human Clinical Trial of the WeFlow-JAAA Endograft System in Patients With Juxtarenal Abdominal Aortic Aneurysms. J Endovasc Ther. 2025 Oct;32(5):1526-1537. doi: 10.1177/15266028231210480. Epub 2023 Nov 24. PMID 37997684